Title: Family Connections: Cultural Adaptation and Feasibility Testing for Rural Latino Communities

NCT number: NCT04731506

Document date: February 6, 2023


#### **CONSENT FORM - SPANISH**

**Título del estudio de investigación** Family Connections

#### Invitación y resumen

Se le invita a estar en este estudio de investigación. La participación en esta investigación es voluntaria. No tiene que participar. Para los propósitos de este documento: Usted puede referirse a:

- Usted mismo/a
- La persona de quien usted es el/la representante legalmente autorizado/a (LAR)
- Su hijo/a menor de 19 años

"Organización" puede referirse a: El Centro Médico de la Universidad de Nebraska (UNMC), Nebraska Medicine (NM), University of Nebraska at Omaha (UNO), o Children s Hospital & Medical Center (CH&MC).

Aquí hay un resumen de la finalidad, los métodos, los riesgos, beneficios y alternativas, para ayudarle a decidir si participar o no en la investigación.

Usted está invitado a participar en este estudio de investigación. La participación en esta investigación es voluntaria. No tienes que participar. A los efectos de este documento: "Usted" puede referirse a:

Usted mismo

La persona de quien usted es el Representante Legalmente Autorizado (LAR) Su hijo menor de 19 años.

"Organización" puede referirse a: University of Nebraska Medical Center (UNMC), Nebraska Medicine (NM), University of Nebraska at Omaha (UNO) o Children's Hospital & Medical Center (CH&MC).

Aquí hay un resumen del propósito, los métodos, riesgos, beneficios y las alternativas, para ayudarlo a decidir si desea o no participar en la investigación.

#### ¿Qué es el programa Family Connections?

Family Connections es un estudio de salud realizado por el Centro Médico de la Universidad de Nebraska (UNMC) en asociación con Central District Health Department - CDHD, Community Action Partnership of Western Nebraska - CAPWN, Two Rivers Public Health department - TRHD, y East Central District Health Department - ECDHD. El estudio comenzó en abril de 2021

En este estudio tenemos un programa de salud para ayudar a las familias a




desarrollar hábitos alimenticios saludables y aumentar la actividad física.

Las personas en este estudio se pondrán en uno de dos grupos. Tienes la misma posibilidad de entrar en cualquiera de los 2 grupos.

#### ¿Qué se me pedirá que haga?

Si acepta ser parte de este estudio, se le pedirá que:

Completar 3 visitas con su hijo(a) (al comienzo del programa, a los 6 meses y 12 meses después del programa) con su trabajador de salud comunitario en un lugar que elija (domicilio o clínica local).

Usar un libro de trabajo.

Completar 2 clases con nuestro entrenador de salud y 10 llamadas telefónicas automatizadas durante un período de 6 meses.

#### ¿Cuáles son los programas?

- Programa A: Las personas en este programa vendrán para su primera visita de estudio con su hijo y completarán 2 visitas con su trabajador de salud comunitario. Esta atención habitual ofrece una opción para estar en una lista de espera para participar en el programa B después de que se complete el estudio.
- Programa B: Las personas en este programa vienen para su primera visita de estudio con su hijo y reciben un libro de trabajo sobre el estilo de vida familiar para llevar a casa. El libro de trabajo ofrece herramientas para ayudar a las familias a comer mejor, ser más activas y controlar el peso. Para ayudar a su familia a mantenerse al día, recibirá 1 llamada de nuestro entrenador de salud y 10 llamadas de soporte automatizadas durante los próximos 6 meses

#### ¿Qué tendré que hacer en cada visita del estudio?

Medimos muchas cosas en cada visita de estudio. Mediremos su presión arterial, cintura, peso y altura. También le pediremos a usted y a su hijo que completen una encuesta. También mediremos la altura y el peso de su hijo. Usted y su hijo(a) recibirán cada uno una tarjeta de regalo de \$25,00, un total de \$50,00 por cada visita de evaluación del estudio (un total de \$150,00 si ambos completan las 3 visitas).

#### ¿Cómo me ayudará el estudio Family Connections?

Puede obtener un programa gratuito para ayudar a su familia a mejorar sus hábitos de vida saludables.

#### ¿Cuáles son los riesgos de participar en el estudio Family Connections?

Los riesgos por participar en el estudio son pequeños. Implican los riesgos normales que tendría por ser más activo.


#### ¿Por qué se le está pidiendo participar en este estudio de investigación?

Se le solicita a usted y a su hijo(a) que participen en este estudio de investigaciónporque se identifica como latino(a) o hispano(a), vive en un área rural, tiene 19 añoso más y tiene un hijo(a) de 6 a 12 años con sobrepeso. u obesidad que vive en suhogar. Si usted está embarazada, amamantando a un bebé o planea quedarembarazada durante este estudio, puede no participar en este estudio.

#### ¿Cuál es la razón para hacer este estudio de investigación?

Este estudio está diseñado para adaptar y probar un programa de salud para ayudar a las familias a desarrollar hábitos alimenticios saludables y aumentar la actividad física. Tanto usted como su hijo han sido invitados a participar en este estudio. El objetivo principal de este programa es mejorar el peso y la salud de usted y su hijo brindándoles consejos útiles para mejorar sus conductas de alimentación y actividad física. El objetivo de este programa es mejorar el peso y la salud de usted y su hijo(a) brindándoles consejos útiles para mejorar sus alimentación y actividad física.

#### ¿Qué se hará durante este estudio de investigación?

Si acepta ser parte de este estudio, usted y su hijo(a) serán colocados en uno de dos grupos. Tienes las mismas posibilidades de entrar en cualquiera de los 2 grupos. ¿Cuáles son los programas?

- Programa A: Las personas en este programa vendrán para su primera visita de estudio con su hijo, completarán 2 visitas con su trabajador de salud comunitario. Esta atención habitual ofrece la opción de estar en una lista de espera para participar en el programa B una vez finalizado el estudio.
- Programa B: Las personas en este programa vienen para su primera visita de estudio con su hijo y reciben un libro de trabajo sobre el estilo de vida familiar para llevar a casa. El libro de trabajo ofrece herramientas para ayudar a las familias a comer mejor, ser más activas y controlar el peso. Para ayudar a su familia a mantenerse al día, recibirá 2 clases de nuestro entrenador de salud y 10 llamadas de soporte automatizadas durante los próximos 6 meses.
- Este estudio incluirá un programa de educación y evaluación de la salud tanto para usted como para su hijo.

#### Evaluación de salud

Como parte de la inscripción en este estudio, usted y su hijo(a) deberán asistir a tresvisitas: una visita de estudio al comienzo del programa, y una visita de estudiodespués de terminar el programa (en aproximadamente 6 meses) y una visita 12meses después de que haya concluido el programa. Las visitas del estudio puedenprogramarse para realizarse en su hogar para su mayor comodidad. La


informaciónde la evaluación de salud de usted y su hijo(a) se recopilará en persona e incluye:

- Encuestas sobre hábitos de alimentación y actividad física, estado de salud, el hogar y la calidad de vida
- Medición de talla, peso y cintura
- Presión arterial

La evaluación de salud de usted y su hijo(a) tomará aproximadamente 30 minutos, ytanto usted como su hijo(a) pueden someterse a las evaluaciones de salud al mismotiempo. Si usted o su hijo(a) no desean efectuar algunas partes de la evaluación desalud o responder a algunas de las preguntas, ni usted ni su hijo(a) están obligadosa hacerlo. En el examen de salud a realizarse durante la visita a los 6 meses, leharemos a usted y a su hijo(a) algunas preguntas sobre lo que les gustó y lo que noles gustó del programa. También se les puede invitar a participar en un grupo focalpara compartir lo que les gustó y lo que no les gustó del programa.

#### Programa de Educación para la Salud Family Connections

Como explicamos antes, usted y su hijo(a) tendrán las mismas posibilidades de ser asignados al grupo A o B. Es posible que se le pida a usted y a su hijo(a) que participen o no en el Programa de Educación para la Salud de Family Connections (programa A). Si usted y su hijo no participan en el Programa de educación sobre la salud de Family Connections, tanto usted como su hijo recibirán la evaluación de salud (descrita anteriormente) en la visita inicial, a los 6 meses cuando complete el programa y después de 12 meses del finalización del programa. Si se les pide a usted y a su hijo(a) que participen en el Programa de educación sobre la salud de Family Connections, este programa comenzará después de que complete su visita inicial y continuará durante 6 meses.

#### Durante este tiempo se le pedirá que:

Complete una llamada telefónica en vivo y complete 10 llamadas telefónicas automatizadas para brindar apoyo y ayudarlos a usted y a su hijo a alcanzar sus objetivos de alimentación y actividad física. La llamada telefónica en vivo tomará aproximadamente 30 minutos y cada llamada automática tomará entre 5 y 10 minutos. Se le pedirá que complete aproximadamente al comienzo del programa una llamada semanal. Eso se reducirá gradualmente a 2 por mes, y una llamada mensual hacia el final.

#### Información de Salud Protegida




Como parte de este estudio, recogeremos información de salud protegida de usted y su hijo(a). La información recogida de usted y su hijo(a) incluirá: edad, raza y etnia, peso y altura corporales, y medicamentos. Como parte de este estudio, la información (incluyendo la información de salud protegida sobre usted y su hijo) recogida durante las llamadas telefónicas que forman parte de este estudio se almacenará inicialmente en una base de datos compatible con HIPPA antes de transferirse al personal de investigación de UNMC. El personal que tendrá acceso a su información y la de su hijo(a) estan listados al final de este formulario.

#### ¿Cuáles son los posibles riesgos de estar en este estudio de investigación?

Hay riesgos mínimos por participar en este estudio. Implican los riesgos normales que tendría por ser más activo. Es posible que el examen de salud pueda causar estrés o ansiedad para usted o su hijo. Usted y su hijo tienen derecho a negarse a participar o a responder cualquier pregunta en el examen de salud. Si usted o su hijo se cansan demasiado durante el examen de salud, pueden tomar un descanso o terminar durante un otro día. También existe un posible riesgo de pérdida de confidencialidad.

#### ¿Cuáles son los posibles beneficios para usted?

Es posible que usted y su hijo(a) no se beneficien de participar en este estudio de investigación. Si usted y su hijo(a) deciden participar en este estudio, no hay garantía de que usted y/o su hijo vean algún cambio en su salud. Sin embargo, usted y/o su hijo(a) pueden recibir los siguientes beneficios: pérdida de peso, aprender a mejorar los comportamientos de alimentación y actividad física y/u otras mejoras en su salud.

#### ¿Cuáles son los posibles beneficios para otras personas?

Es posible que la información obtenida de este estudio pueda ayudar a desarrollar programas que puedan usarse para alentar a las familias hispanas y latinas a llevar un estilo de vida más activo y saludable.

#### ¿Cuáles son las alternativas para estar en este estudio de investigación?

En lugar de participar en este estudio de investigación, puede optar por no participar y continuar con la atención estándar en su clínica comunitaria y/o departamento de salud local.

#### ¿Cuánto le costará estar en este estudio de investigación?

No hay ningún costo para usted o su hijo(a) por participar en este estudio de investigación.


#### ¿Se le pagará a usted por estar en este estudio de investigación?

Usted y su hijo(a) recibirán una compensación por su participación en este estudio de investigación. Usted y su hijo(a) recibirán su compensación del estudio al finalizar cada visita requerida por el estudio.

Recibirá \$25 y su hijo recibirá \$25 en cada visita (un total de \$50 por cada visita). Esto se suma a un total de \$ 150 si ambos completan las 3 visitas.

#### ¿Quién está pagando por esta investigación?

Los National Institutes of Health (NIH) nos dan dinero para hacer investigaciones como este estudio.

## ¿Qué debe hacer si se lesiona o tiene un problema médico durante este estudio de investigación?

Su bienestar y el de su hijo(a) es la principal preocupación de todos los miembros del equipo de investigación. Si usted o su hijo(a) tienen un problema como resultado directo de participar en este estudio, debe ponerse en contacto de inmediato con una de las personas listadas al final de este formulario de consentimiento.

#### ¿Cómo se protegerá la información sobre usted?

Usted y su hijo(a) tienen derechos con respecto a la protección y privacidad de la información médica recopilada antes y durante esta investigación. Esta información médica se denomina "información de salud protegida" (PHI, por sus siglas en inglés). La PHI utilizada en este estudio puede incluir la dirección, fecha de nacimiento, historial médico, los resultados de los exámenes físicos, así como los resultados de otros procedimientos de investigación de usted y de su hijo(a). Solo se recopilará la cantidad mínima de PHI para esta investigación. Los registros médicos y de investigación de su hijo(a) se conservarán de manera segura. En el futuro, podemos eliminar los identificadores de la información. Es posible que esta información anonimizada pueda ser utilizada para otras investigaciones por nosotros o por otro investigador, sin pedir su permiso.

#### ¿Quién tendrá acceso a la información sobre usted?

Al firmar este formulario de consentimiento, nos permite (a los investigadores enumerados en este formulario de consentimiento y a otras personas involucradas en esta investigación en la Organización) tener acceso a sus datos de investigación. Los datos de su investigación se utilizarán únicamente para los fines descritos en la sección ¿Cuál es la razón para hacer este estudio de investigación?

Puede cambiar de opinión y pedirnos que dejemos de recopilar más datos de investigación para utilizarlos en esta investigación en cualquier momento. Puede


ponerse en contacto con el investigador principal o cualquiera de los miembros del personal del estudio que figuran al final del formulario de consentimiento. Sin embargo, la información que se incluye en los datos de investigación obtenidos hasta la fecha aún se puedeutilizar. Si cancela esta autorización, ya no podrá participar en esta investigación.

Es posible que compartamos sus datos de investigación con otros grupos:

- La Junta de Revisión Institucional (IRB) de UNMC
- Funcionarios institucionales designados por el UNMC IRB
- La Oficina para la Protección de Seres Humanos en Estudios de Investigación (OHRP, en inglés) del Departamento de Salud y Servicios Humanos de los Estados Unidos (HHS, en inglés)
- Institutos Nacionales de Salud (NIH)
- Above Ground Development (una empresa que cumple con HIPPA contratada para realizar las llamadas telefónicas automatizadas)

Usted nos permite usar y compartir sus datos de investigación y los de su hijo(a) durante el tiempo que dure la investigación.

### ¿Cómo se pondrán a su disposición los resultados de la investigación durante y después de que finalice el estudio?

La información obtenida durante la investigación que no se compartirá con usted son los resultados generales o parciales del programa en el que participará. Los resultados individuales suyos y de su hijo se compartirán con usted. Al firmar esta autorización, renuncia temporalmente a su derecho a ver esta información relacionada con la investigación mientras se lleva a cabo la investigación. Podrá ver esta información si lo desea después de que se complete la investigación.

En la mayoría de los casos, los resultados de la investigación pueden estar disponibles para usted cuando se completa el estudio y el investigador revisa todos los resultados. La información de este estudio puede publicarse en revistas científicas o presentarse en reuniones científicas, pero su identidad y la de su hijo se mantendrán estrictamente confidenciales.

Si desea los resultados del estudio, comuníquese con la Investigadora Principal al número de teléfono que aparece al final de este formulario o escribiendo a la Investigadora Principal a la siguiente dirección:

Dra. Fabiana Brito Silva 984365 Nebraska Medical Center

IRBVersion 1


Omaha, NE 68198-4365

Una descripción de este ensayo clínico estará disponible en el sitio www.ClinicalTrials.gov, según lo exige la ley de EE. UU. Este sitio no incluirá información que pueda identificarlo. A lo sumo, el sitio incluirá un resumen de los resultados. Puede buscar este sitio en cualquier momento.

#### ¿Qué pasará si decide no participar en este estudio de investigación?

Puede decidir no participar en este estudio de investigación. Decidir no participar en esta investigación no afectará su relación con el investigador o la organización. No perderá ningún beneficio al que tenga derecho.

#### ¿Qué pasará si usted decide dejar de participar una vez que comience?

Puede dejar de participar en esta investigación (retirarse) en cualquier momento. Simplemente llame al investigador o a cualquier miembro del personal de investigación.

La decisión de retirarse no afectará su cuidado de la salud ni su relación con el investigador o esta institución. No perderá ningún beneficio al que tenga derecho.

Puede decidir no dar permiso para que su hijo(a) participe en este estudio de investigación, o puede detener su participación en este estudio de investigación ("retirarse") en cualquier momento antes, durante o después de que comience la investigación. Decidir no participar en este estudio de investigación o decidir retirarse no afectará la relación de su hijo(a) con el investigador o la Institución. Su hijo(a) no perderá ningún beneficio al que tenga derecho.

Usted y su hijo(a) pueden ser retirados del estudio si no sigue las instrucciones del investigador o del equipo de investigación.

Usted y su hijo también pueden ser retirados del estudio si:

- Usted y su hijo(a) no asisten a las visitas de estudio requeridas
- No completa las llamadas telefónicas de estudio requeridas

#### ¿Se le dará alguna información importante durante el estudio?

Le informaremos de inmediato si recibimos nueva información que pueda hacerle cambiar de opinión sobre la participación de usted y su hijo en el estudio.

#### ¿Qué debe hacer si tiene alguna pregunta sobre el estudio?

Se le ha entregado una copia del folleto "¿Qué debo saber antes de participar en un

IRBVersion 1


estudio de investigación?" Si tiene alguna pregunta en cualquier momento sobre este estudio, debe comunicarse con el investigador principal o con cualquiera de los miembros del personal del estudio que figuran en este formulario de consentimiento o en cualquier otro documento que se le entregue.

#### ¿Cuáles son sus derechos como participante de investigación?

Usted y su hijo(a) tienen derechos como sujetos de investigación. Estos derechos sehan explicado en este formulario de consentimiento y en el material Los Derechos delos Sujetos de Investigación que se le ha entregado. Si tiene alguna pregunta sobreestos derechos o quejas sobre la investigación, puede comunicarse con cualquierade las siguientes personas:

- El investigador u otro personal del estudio, o la Junta de Revisión Institucional (IRB)
- Teléfono: (402) 559-6463. Correo electrónico: IRBORA@unmc.edu
- Por correo: Junta de Revisión Institucional de UNMC, 987830 Nebraska Medical Center, Omaha, NE 68198-7830
- Defensor del Sujeto de Investigación al Teléfono: (402) 559-6941
- Correo electrónico: unmcrsa@unmc.edu

#### Documentación del consentimiento informado

Usted toma libremente la decisión de dar permiso para que su hijo(a) participe en este estudio de investigación. Firmar este formulario significa que:

- Ha leído y comprendido este formulario de consentimiento.
- Le han explicado el formulario de consentimiento.
- Se le ha entregado una copia de Los Derechos de los Sujetos de Investigación
- Ha obtenido respuesta a sus preguntas
- Ha decidido permitir que su hijo(a) participe en el estudio de investigación.
- Le han dicho que puede hablar con uno de los investigadores que se enumeran a continuación en este formulario de consentimiento si tiene alguna pregunta durante el estudio.
- Se le entregará una copia firmada y fechada de este formulario de consentimiento para que la conserve.

Cláusula de consentimiento del niñoSi se invita a su hijo(a) a participar en este estudio, usted se registra para dar su permiso. Cada niño puede aceptar participar en un estudio a su propio nivel de comprensión. Cuando firma este formulario, también indica que su hijo(a) comprende y acepta participar en este estudio según su comprensión.




| Firma del Sujeto | Fecha_ | |
|---|---|---|
| Firma de la madre/padre | | Fecha |
| Mi firma certifica que | todos los elemen | tos del consentimiento |
| informado | descritos | en |
| este formulario de cons | entimiento han si | do explicados completa |
| mente al | sujeto. | A mi |
| juicio, el sujeto posee la capacidad legal para dar su consent | | |
| imiento | informado | para |
| participar en esta inve | stigación y está | voluntariamente y con |
| conocimiento | de | causa |
| dando | su | con |
| sentimiento | informado | pa |
| ra participar.Firma | de la persor | na que obtiene el |
| consentimiento | | <u></u> |
| Fetcha | | |

#### Personal autorizado del estudio:

#### Principal

\* Silva, Fabiana (Fabiana) alt #: 402-552-6363

degree: PhD

#### Secondary

\* Almeida, Fabio

phone: 402-559-9395 alt #: 402-559-9395

degree: PhD

#### **Participating Personnel**

\* Ochoa-Rojas, Daisy phone: 402-559-4325 alt #: 402-552-6363

degree: BS

\* Santos, Natalia phone: 402-559-4325 alt #: 402-305-5315 degree: MPH

## ¿Qué Necesito Saber Antes De Participar En Un Estudio De Investigación?

Usted ha sido invitado a participar en un **estudio de investigación**. Los estudios de investigación también se conocen como pruebas clínicas o protocolos. **La investigación** es un plan organizado diseñado para obtener nuevos conocimientos sobre una enfermedad o la función normal del cuerpo. A las personas que participan en una investigación se les llama **sujetos de investigación**. **El investigador** es la persona a cargo del estudio de investigación. Usted recibirá información del investigador y el equipo de investigación, y luego se le pedirá que ofrezca su consentimiento para participar en la investigación.

Esta hoja le servirá para pensar sobre preguntas que le hará al investigador o a su personal. Usted deberá conocer <u>todas</u> estás respuestas antes de decidir participar en la investigación.

- ¿Cuál es el **propósito** de la investigación? ¿Por qué el investigador está haciendo la investigación?
- ¿Cuáles son los riesgos de la investigación? ¿Qué cosas malas podrían ocurrir?
- ¿Cuáles son los posibles **beneficios** de la investigación? ¿Cómo podría ayudarme esto?
- ¿Cuán diferente es esta investigación del cuidado o tratamiento que recibiría si no estuviera participando de ella? ¿Existen otros tratamientos que yo pueda recibir?
- ¿Reciben **todos** los participantes en este estudio el mismo tratamiento?
- ¿Me cuesta algo adicional participar en esta investigación?
- ¿Tengo que participar de esta investigación? ¿Recibiré cuidado de mi médico aún cuando diga que no?
- ¿Puedo retirarme de la investigación una vez comience? ¿Cómo?
- ¿Quién tendrá acceso a mis expedientes?
- ¿Cómo contacto al investigador si tengo más preguntas?
- ¿A quién llamo si tengo preguntas sobre mi participación como **sujeto de investigación**?

Asegúrese de que todas sus preguntas son contestadas antes de que decida si participa o no en la investigación.

# LOS DERECHOS DE LOS PARTICIPANTES DE INVESTIGACIÓNES COMO PARTICIPANTE EN UNA INVESTIGACIÓN EN EL CENTRO MEDICO DE NEBRASKA USTED TIENE EL DERECHO

de ser informado de todo lo que necesita saber referente a la investigación antes de que se le pida decidir si desea participar en la investigación. Los detalles de la investigación se le serán expilcado de un manera que asegure que Usted los entienda suficientmente para decidir si quiere o no participar en la investigación.

de decidir libremente si quiere participar en la investigación.

de decidir no participar en la investigación o de dejar de participar en la investigación en qualqier momento. Esto no afectará su relación con el investigador, la Universidad de Nebraska o el Centro Médico de Nebraska. Si Usted se encuentra participando en una investigación, la decisión de dejar de participar en la investigación no afectará a sus cuidados médicos y su médico seguirá atendiendlo.

de hacer preguntas acerca de la investigación cuando Usted lo desea. El investigador le contestará sus preguntas de una manera honesta y completa.

saber que su seguridad y bienestar siempre seran de primera importancia. El investigador demostrará el grado más alto de abilidad y cuidado hacia el paciente durante la investigación. Los riesgos y las molestias asociadas con la investigación seran minimizados lo máximo que sea posible.

a privacidad and confidencialidad. El investigador tratará sus datos personales con cuidado y respetará su confidencialidad.

... de mantener los derechos legales que ahora tiene. Al participar en esta investigación Usted no esta cediendo sus derechos legales.

de ser siempre tratado con dignidad y con respeto

El Comité Institucional De Revisión de Investigaciones es responsible de asegurar que sus derechos y bienestar son protejidos. Si Usted tiene preguntas sobre sus derechos, comuníquese con El Comité Institucional De Revisión de Investigaciones al (402) 559-6463.